CLINICAL TRIAL: NCT00719498
Title: Early High-dose Erythropoietin Therapy and Hypothermia After Out-of-hospital Cardiac Arrest: A Matched Control Study
Brief Title: Effect of Early High-dose Epoetin Alfa During Cardiac Arrest (Pilot Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Cilag S.A.S. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005008
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Resuscitation; Cardiopulmonary; Cardiac Arrest
Keywords: Epo-alpha; Cardiac arrest; Mild hypothermia
MeSH Terms: conditions — Heart Arrest

INTERVENTIONS:
Drug: Epo-alpha

SUMMARY:
The purpose of this study is to test the possible neuroprotective effect of early high dose erythropoietin alpha after out of hospital cardiac arrest (OHCA).

DETAILED DESCRIPTION:
Aim: To test the possible neuroprotective effect of early high-dose erythropoietin alpha after out-of-hospital cardiac arrest (OHCA). Safety, pharmacokinetics and an estimation of potential risks benefits of EPO treatment were evaluated. Methodology: An open labelled, pilot, matched control study. Following resuscitation with mild hypothermia with after OHCA, participants received a first dose of EPO-alpha followed by four additional injections within 48 hours (40 000 IU intravenously each injection). Plasma Epo-alpha levels were measured at different time points. Outcome and adverse events were assessed up to day 28 and were compared with those of matched-paired controls Pilot, open-labelled, matched controls study performed between Nov 2003 and May 2004. As the first step, the effect of high-dose Epo-alpha for 20 consecutive patients with OHCA who had been successfully resuscitated by the emergency medical service was studied. The participants received the first dose of Epo-alpha as soon as possible after stable ROSC, followed by an additional injection every 12h during the first 48 hours ICU admission (40 000 IU intravenously each injection). Collected data included demographics, clinical characteristics, biological features, treatment and outcome. Severity was assessed by the Simplified Acute Physiologic Score 2 (SAPS2). Mortality and neurological outcome were recorded at day 28. All unexpected events were assessed in order to detect potential side effects of High-dose Epo administration. As the second step, the outcomes observed among the prospective Epo-treated patients were compared to the cohort with outcomes observed among case-matched historical controls. Two matched controls were selected for each Epo-treated patient. Neurological assessment was performed on admission and each day between days 1 and 7, and at days 14, 21 and 28. Blood samples were drawn daily from day 1 to day 7 and weekly from day 7 to day 28. For the pharmacokinetics blood samples were drawn just before and at 2h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 78h, 84h, and 96 h after the first administration of Epo-alpha.

Intravenous Epo-alpha: First dose as soon as possible after stable return of spontaneous circulation (ROSC), followed by an additional injection every 12 hours during the first 48 hours. (40 000 IU at each injection)

ELIGIBILITY:
Inclusion Criteria:

* Patients who have OHCA of presumed cardiac origin
* Patient's who have delay between the collapse and onset of cardiopulmonary resuscitation (CPR, no flow) less that 10 minutes
* Patient's who have delay between onset of CPR and return of spontaneous circulation (ROSC, low flow) less than 50 minutes
* Patient's who have persistent coma with Glasgow Coma Scale (CGS) less that 7 after ROSC

Exclusion Criteria:

* Patient's who have cardiac arrest of non-cardiac aetiology
* Patient who have previous EPO treatment
* Patient's who are in pregnancy stage
* Patient's who have evidence of rapidly fatal underlying condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-11; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Primary: Mortality and neurological outcome recorded at day 28

SECONDARY OUTCOMES:
All unexpected events in order to detect potential side effects of High-dose Epo administration

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A.S. Clinical Trial, Study Director — Janssen Cilag S.A.S.

REFERENCES:
- [Result] Cariou A, Claessens YE, Pene F, Marx JS, Spaulding C, Hababou C, Casadevall N, Mira JP, Carli P, Hermine O. Early high-dose erythropoietin therapy and hypothermia after out-of-hospital cardiac arrest: a matched control study. Resuscitation. 2008 Mar;76(3):397-404. doi: 10.1016/j.resuscitation.2007.10.003. Epub 2007 Nov 26. PMID 18037223
- See also: Effect of early high-dose Epoetin alfa during cardiac arrest (pilot study) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=274&filename=CR005008_ScienceDirect.pdf